CLINICAL TRIAL: NCT05441566
Title: Dynamic Monitoring and Significance of Molecular Residual Disease After Surgery in Driver Gene-positive and Driver Gene-negative Stage IB-IIA NSCLC
Brief Title: Significance of MRD After Surgery in Driver Gene-positive and Driver Gene-negative Stage IB-IIA NSCLC
Status: Enrolling by invitation | Type: Observational
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ShenzhenPH 0606
Record Dates: First submitted 2022-06-16; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: NSCLC MRD ctDNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Driver gene-positive
- Driver gene-negative

SUMMARY:
1. It has been controversial whether adjuvant therapy should be done for patients with stage IB NSCLC after surgery in clinical practice, and identifying patients with high-risk recurrence and those who can benefit from adjuvant therapy is an important clinical problem to be solved. Therefore, the first key scientific issue to be solved in this topic is to analyze the correlation between MRD detection results and both recurrence and adjuvant therapy efficacy by focusing on the stage IB-IIA postoperative NSCLC patient population. To provide clinical data to aid clinical screening of NSCLC patients at high risk of recurrence after surgery in stage IB-IIA.

2, if the detection of MRD has important clinical value such as accurately identifying the population at high risk of recurrence of stage IB-IIA NSCLC, the differences in MRD, etc. between driver gene-positive and -negative patients require further comparative analysis. The second key scientific issue to be solved in this topic is: the different role of MRD in driver gene-positive and driver gene-negative patients: comparison of positive rates, analysis of prognostic differences; and providing clinical data for elucidating the differences between driver gene-positive and -negative patients in MRD evaluation of lung cancer.

3. If MRD is different between NSCLC patients with positive and negative driver genes in stage IB-IIA, is there a difference in the biological behavior of the tumors themselves between these two types of patients? Is there a difference in the ability of the tumor tissue itself to shed tumor cells to be released into the blood? The third scientific question to be addressed in this project is to explore the difference in the ability of patients with stage IB-IIA NSCLC to release ctDNA from their tumors by analyzing the correlation between detailed clinicopathological data and MRD. To provide a scientific basis for exploring the differences in tumor biological behavior between NSCLC driver gene positive and negative.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage I-II operable NSCLC in AJCC TNM stage (8th edition) confirmed by clinical pathological staging;
2. The physical condition and organ function allow surgery and postoperative adjuvant therapy；
3. At the time of signing the informed consent form, the age is equal to or greater than 18 years old;
4. Tumor histology or cytology confirmed NSCLC;
5. Never received any surgery, radiotherapy, chemotherapy or molecular targeted anti-tumor therapy;
6. Eastern Cooperative Oncology Group performance status score (ECOG PS) is 0 ~ 1 points;
7. Patients agree and have the ability to follow the planned study visits, treatment plan, laboratory tests and other research steps;
8. Expected survival time ≥ 6 months.

Exclusion Criteria:

1. Patients with other malignant tumors;
2. Patients with inoperable clinical evaluation;
3. Patients with other serious diseases that may affect follow-up and significant short-term survival;
4. Patients who have received previous anti-tumor treatment such as surgery, chemotherapy, targeted or immunotherapy;
5. Eastern Cooperative Oncology Group performance status score (ECOG PS) > 2 points;
6. Patients with clinically clear active infection, including but not limited to pneumonia;
7. Any other condition and social/psychological problems, etc., judged by the investigator that the patient is not suitable for participating in this study; can not accept the use of contrast-enhanced magnetic resonance imaging (MRI) or contrast-enhanced computed tomography (CT) for clinical follow-up;
8. Other researchers think it is not suitable;
9. or can not comply with the study protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is an open-label, single-center study to explore the clinical significance of MRD in Chinese adult patients with operable stage I-II lung cancer with positive and negative driver gene mutations of NSCLC. The study will include 60 patients with stage I-II NSCLC who are treated surgically in our center.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in ctDNA levels after surgery 2 years | baseline and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gui G Ding, Principal Investigator — Shenzhen People's Hospital
Locations (1):
- ShenzhenPH, Shenzhen, China